CLINICAL TRIAL: NCT05793268
Title: Safety and Efficacy of Finite Versus Continuous Nucleos(t)Ide Analogues Therapy in Patients With Chronic Hepatitis B: A Multicenter Randomized Controlled Trial
Brief Title: Finite Versus Continuous Nucleos(t)Ide Analogues for Chronic Hepatitis B
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Yao-Chun Hsu, Professor, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMRP26111N
Record Dates: First submitted 2022-12-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis b
Keywords: hepatitis b virus infection; antiviral therapy; randomized trial
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finite Therapy (Experimental): Discontinuation of nucleos(t)ide analog (Nuc) therapy
  Interventions: Other: Nuc Discontinuation
- Continuous Therapy (Active Comparator): Continuation of oral Nuc monotherapy using entecavir (0.5mg/tab, once per day), tenofovir disoproxil fumarate (300mg/tab, once per day), or tenofovir alafenamide (25mg/tab, once per day) for 3 years
  Interventions: Drug: Entecavir or Tenofovir

INTERVENTIONS:
Other: Nuc Discontinuation — Eligible patients are randomly allocated with a 1:1 ratio to continue viral suppression or stop the treatment (entecavir or tenofovir). Patients will be followed up for 3 years. For patients who are assigned to the finite Nuc therapy, they should be monitored monthly for the initial 3 months and then every 3-6 months thereafter for relapse.
  Arms: Finite Therapy
Drug: Entecavir or Tenofovir — Continuation of either entecavir or tenofovir treatment for 3 years
  Arms: Continuous Therapy

SUMMARY:
BACKGROUND:

Finite nucleos(t)ide analogue (Nuc) therapy was proposed as an alternative strategy in the management of chronic hepatitis B (CHB) but there remained not data from randomized controlled trials to clarify safety and efficacy of this treatment strategy.

AIMS:

The investigators aimed to evaluate the safety and efficacy of finite Nuc therapy versus continuous treatment in CHB patients without liver cirrhosis and also to identify factors that may predict therapeutic responses and clinical outcomes after withdrawal of Nuc treatment for CHB

MATERIAL AND METHODS:

This is a multicenter randomized controlled trial conducted in Taiwan. Eligible patients are adults (age≥20 years) with CHB (chronic infection ≥ 6 months) who fulfill the APASL guideline 2016 to stop NA therapy. Those with cirrhosis, malignancy, organ transplant, autoimmune disorder, or serious underlying diseases including renal impairment were excluded. A total of 360 patients will be enrolled. Enrolled patients are randomly allocated with a 1:1 ratio to continue viral suppression with entecavir (0.5mg once daily) or tenofovir disoproxil fumarate (300mg once daily) or stop the treatment. All patients will be followed up according to the protocol recommended by a panel of APASL experts. The primary analysis for study outcomes is scheduled at 3 years after randomization and the primary outcome is seroclearance of HBsAg. There will be interim analyses scheduled at one- and two-years following randomization of the first 200 patients, and also one-and two years following randomization of the planned 360 patients, to determine whether early termination of the trial may be justified by attainment of the efficacy endpoint (10% vs 1% of HBsAg seroclearance) or concerns of the safety outcomes (significant between-group difference in mortality, acute on chronic liver failure, or acute flares with hepatic decompensation).

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection imposes a serious threat to global public health, affecting more than 250 million individuals around the world. In the management of patients with chronic hepatitis B (CHB), treatment with nucleos(t)ide analog (Nuc) has been shown to improve clinical outcomes including occurrence and recurrence of hepatocellular carcinoma (HCC), liver-related mortality, and overall mortality. Nuc therapy, however, cannot exterminate HBV and so continuous treatment is usually required to sustain viral inhibition. Seroclearance of hepatitis B surface antigen (HBsAg) predicts durable remission off Nuc and may serve as the treatment endpoint, but it rarely occurs with current regimen. Therefore, long-term to indefinite treatment is currently recommended.

In view of various concerns such as drug exposure, adherence, and expense for a treatment course that could be lifelong, a finite strategy of Nuc therapy was proposed to allow treatment withdrawal prior to HBsAg seroclearance. Another major reason for the finite strategy is a higher chance of HBsAg seroclearance following treatment cessation. Nevertheless, viral replication almost always reactivates and often leads to clinical flares. While an episode of acute flare might be self-limited or even conducive to HBsAg seroclearance, it could progress to acute on chronic liver failure with fatal consequences. Risks of these serious outcomes following treatment withdrawal need to be accurately quantified in order to inform the practice of finite Nuc therapy.

Existent literature on the efficacy and safety of finite Nuc therapy remained very limited, as recently shown in a systematic review and meta-analysis by Hall and colleagues. In order to close the gaps in current knowledge, the investigators conduct this multicenter randomized controlled trial to examine if cessation of Nuc is safe and conducive to HBsAg seroclearance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Chronic hepatitis B virus infection (defined as positive HBsAg for ≥ 6 months)
3. Entecavir or tenofovir (either tenofovir disoproxil fumarate or tenofovir alafenamide) for at least two years and still on therapy at screening for this trial.
4. Fulfillment of the stopping rules recommended by the Asian-Pacific guidelines 2016:

   * For patients with positive HBeAg prior to their antiviral treatment, HBeAg seroconversion needs to be documented and followed by consolidation treatment for at least one year). Besides, serum ALT is within normal limits and HBV DNA is undetectable.
   * For those with negative HBeAg prior to the antiviral therapy, undetectable HBV DNA documented on three separate occasions (at least 6 months apart)
5. At screening for this study, HBsAg serology is positive, HBeAg negative, and HBV DNA undetectable in serum.

Exclusion Criteria:

1. Liver cirrhosis (either clinical or pathological diagnosis) at screening
2. Serious underlying disease (with valid certification of catastrophic illness) at screening
3. Manifestations and concerns of hepatic decompensation, including serum bilirubin >2mg/dL and/or prolongation of prothrombin time > 3 seconds at screening
4. Hepatitis C virus (if anti-HCV serology is positive, confirmation with detectable HCV RNA is required), human immunodeficiency virus (HIV) or hepatitis delta virus (HDV) coinfection at screening.
5. Prior history of any malignancy including liver cancer
6. Prior history of any organ transplantation
7. Prior history of drug resistance to any Nuc agent
8. Any patient condition that the treating physician deems inappropriate for enrollment in this trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with seroclearance of HBsAg | The time from randomization to seroclearance of HBsAg, up to 3 years after randomization
  Serology of HBsAg was negative by the laboratory report

SECONDARY OUTCOMES:
Number of Participants with liver-related mortality or liver transplantation | The time from randomization to this secondary outcome, up to 3 years after randomization
  Death from liver failure or liver transplantation because of liver failure
Number of Participants with acute on chronic liver failure | The time from randomization to this secondary outcome, up to 3 years after randomization
  According to the definition of Asian-Pacific Association for the Study of Liver Diseases
Number of Participants with severe acute exacerbation of chronic hepatitis B | The time from randomization to this secondary outcome, up to 3 years after randomization
  Serum alanine aminotransferase > 5 times the upper limit of normal with either serum bilirubin ≥2mg/dL or prolongation of prothrombin time ≥3 seconds, in the presence of serum HBV DNA >2000 IU/mL
Number of Participants with clinical relapse of active hepatitis B | The time from randomization to this secondary outcome, up to 3 years after randomization
  Serum alanine aminotransferase > 2 times the upper limit of normal in the presence of serum HBV DNA >2000 IU/mL
Number of Participants with incident hepatocellular carcinoma | The time from randomization to this secondary outcome, up to 3 years after randomization
  Diagnosis of hepatocellular carcinoma after randomization
Changes in the FIB4 index from baseline | At three years after randomization
  The formula for FIB-4 is: Age ([yr] x AST [U/L]) / ((PLT [10(9)/L]) x (ALT [U/L])(1/2)).
Changes in serum concentration of quantitative HBsAg from the baseline at randomization | At three years after randomization
  Quantitative HBsAg measured in log IU/mL
Changes in serum concentration of HBcrAg from the baseline at randomization | At three years after randomization
  Quantitative HBcrAg measured in log U/mL
Changes in the quality of life as measured by Short Form-36 Inventory from the baseline | At each follow-up visit during the study period, up to 3 years after randomization
  Chinese version of the Short-form 36. Responses in each domain are transformed into a 0-100 scale, with a higher score indicating better health or functioning.
Changes in the scores measured by the General Anxiety Disorder-7 from baseline | At each follow-up visit during the study period, up to 3 years after randomization
  Chinese version of the questionnaire. The total score can range from 0 to 21, with a higher score indicating more severe anxiety
Direct expenditure on healthcare | At three years after randomization
  Money (measured in US dollars) that is paid for all sort of healthcare
Changes in the scores measured by the Perceived Stress Scale - 14 from baseline | At each follow-up visit during the study period, up to 3 years after randomization
  Chinese version of the questionnaire. The total score can range from 0 to 56, with a higher score indicating a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chun Hsu, MD, PhD, Principal Investigator — E-Da Hospital/I-Shou University
Locations (6):
- Taiwan (6):
  - Chia-Yi Christian Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Fu-Jen Catholic University Hospital, Taipei
  - Taitung Mackay Memorial Hospital, Taitung
  - Lotung Poh-Ai Hospital, Yilan

IPD SHARING:
Plan to Share IPD: Yes
Data collected during this trial, including de-identified individual participant data and data dictionaries defining fields in the datasets will be available to access. Documents that include the study protocol, statistical analysis plan, and informed consent form will also be available. Data access will be provided to investigators for academic research after a proposal has been approved by the study committee identified for this purpose. The investigator will sign a data access agreement on how to collaborate with consideration of potential overlaps between the proposal and ongoing efforts. Data will be available beginning with full publication of this Article. Proposals should be directed to the Principal Investigator (Dr. Yao-Chun Hsu), and the de-identified database will be transferred by email.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available beginning with full publication of the study results in an academic peer-reviewed journal and for at least a year.

REFERENCES:
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Kao JH, Jeng WJ, Ning Q, Su TH, Tseng TC, Ueno Y, Yuen MF. APASL guidance on stopping nucleos(t)ide analogues in chronic hepatitis B patients. Hepatol Int. 2021 Aug;15(4):833-851. doi: 10.1007/s12072-021-10223-5. Epub 2021 Jul 23. PMID 34297329
- [Background] Hsu YC, Yeh ML, Wong GL, Chen CH, Peng CY, Buti M, Enomoto M, Xie Q, Trinh H, Preda C, Liu L, Cheung KS, Yeo YH, Hoang J, Huang CF, Riveiro-Barciela M, Kozuka R, Istratescu D, Tsai PC, Accarino EV, Lee DH, Wu JL, Huang JF, Dai CY, Cheung R, Chuang WL, Yuen MF, Wong VW, Yu ML, Nguyen MH. Incidences and Determinants of Functional Cure During Entecavir or Tenofovir Disoproxil Fumarate for Chronic Hepatitis B. J Infect Dis. 2021 Dec 1;224(11):1890-1899. doi: 10.1093/infdis/jiab241. PMID 33999179
- [Background] Berg T, Simon KG, Mauss S, Schott E, Heyne R, Klass DM, Eisenbach C, Welzel TM, Zachoval R, Felten G, Schulze-Zur-Wiesch J, Cornberg M, Op den Brouw ML, Jump B, Reiser H, Gallo L, Warger T, Petersen J; FINITE CHB study investigators [First investigation in stopping TDF treatment after long-term virological suppression in HBeAg-negative chronic hepatitis B]. Long-term response after stopping tenofovir disoproxil fumarate in non-cirrhotic HBeAg-negative patients - FINITE study. J Hepatol. 2017 Nov;67(5):918-924. doi: 10.1016/j.jhep.2017.07.012. Epub 2017 Jul 21. PMID 28736139
- [Background] Jeng WJ, Chen YC, Chien RN, Sheen IS, Liaw YF. Incidence and predictors of hepatitis B surface antigen seroclearance after cessation of nucleos(t)ide analogue therapy in hepatitis B e antigen-negative chronic hepatitis B. Hepatology. 2018 Aug;68(2):425-434. doi: 10.1002/hep.29640. Epub 2018 May 6. PMID 29108132
- [Background] Hall SAL, Vogrin S, Wawryk O, Burns GS, Visvanathan K, Sundararajan V, Thompson A. Discontinuation of nucleot(s)ide analogue therapy in HBeAg-negative chronic hepatitis B: a meta-analysis. Gut. 2022 Aug;71(8):1629-1641. doi: 10.1136/gutjnl-2020-323979. Epub 2021 Sep 7. PMID 34493592